CLINICAL TRIAL: NCT06797102
Title: Comparative Effects of Neuromuscular Training Vs Close Chain Exercises in Athletes With Post Operative ACL Injury
Acronym: NMTvsCC-ACL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0423
Record Dates: First submitted 2025-01-10; First posted 2025-01-28 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Sports Physical Therapy
Keywords: acl; neuromuscular exercises; close chain exercises; pain; range of motion; strength; endurance; athletes; post operative
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A neuromuscular training (Experimental): Patients in this group received a neuromuscular training protocol along with general treatment for 10 minutes
  Interventions: Other: Neuromuscular Exercises
- Group B Close chain exercises (Experimental): Patients in this group will receive close chain exercises for core strengthening along with general treatment for 10 min
  Interventions: Other: Close Chain Exercises

INTERVENTIONS:
Other: Neuromuscular Exercises — Patients in this group received a neuromuscular training protocol along with general treatment for 10 minutes. This included hot packs, lumbar stretches, and ergonomic posture correction divided over 6 weeks The exercises performed included squatting, single leg stance, and balance reach leg and arm exercises with 10 repetitions each. They also did lunge exercises with five repetitions bilaterally, step up and down exercises with 10 repetitions, single leg standing on a balance mat with 10 repetitions and a 10-second hold, single board exercises, and single leg stance with weights and eyes closed for five minutes with a 10-second hold. Additionally, they stood on a wobble board with eyes closed five times with a 10-second hold. The protocol included running on a treadmill and trampoline for five minutes per day, running figure-of-eight patterns, and agility drills at a slow speed for five minutes each.
  Arms: Group A neuromuscular training
Other: Close Chain Exercises — Patients in this group received closed chain exercises for core strengthening along with general treatment for 10 minutes, including hot packs, lumbar stretches, and ergonomic posture correction, divided over 6 weeks. The exercises included sets of squats, lunges, leg presses, wall squats, standing heel raises on a single leg, and single leg dead lifts. Each treatment session lasted 60 minutes, incorporating a warm-up and cool-down period of 10 minutes.
  Arms: Group B Close chain exercises

SUMMARY:
The aim of this study is to determine the effects of close chain exercises and neuromuscular training on pain, range of motion, strength and endurance in athletes with post operative ACL injury The study will be randomized control trial with the sample size of 36. Subjects will be enrolled according to inclusion and exclusion criteria. Patients will be divided into two groups, each with 18 patients. Group A will receive Neuromuscular training while Group B will receive Close chain exercises. The participants will receive treatment sessions over 6-week period. The treatment session will be of 60 minutes with a warm up and cool down period of 10 minutes. Outcome measures in both groups will be assessed by International Knee Documentation Committee Evaluation Form. Score for function, Numeric Pain Rating Scale (NPRS) for pain, Goniometer to measure range of motion, single leg hop, squats, triple jump test, push ups for strength and endurance respectively.

DETAILED DESCRIPTION:
Objective of my study is to compare the effects of Neuromuscular Training vs Close Chain Exercises on pain, range of motion, strength and endurance in athletes with post operative ACL injury

ELIGIBILITY:
Inclusion Criteria:

* Athletes aged 18 to 35 years
* 6-9 months after ACL reconstruction
* Athletes who sustained unilateral ACL injury treated surgically
* Athletes returning to sports
* minimal to no knee effusion
* normal knee range of motion
* Willing to take post-operative exercise program

Exclusion Criteria:

* History of lower extremity fractures surgery or traumatic injuries
* Neuromuscular disease
* Systemic disease
* Patients who had history of prior knee surgery were excluded

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Male
Enrollment: 36 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
International Knee Documentation Committee (IKDC) Subjective Knee Form | 6 months
  The IKDC Questionnaire is a subjective scale that provides patients with an overall function score. The questionnaire looks at 3 categories: symptoms, sports activity, and knee function. The symptoms subscale helps to evaluate things such as pain, stiffness, swelling and giving-way of the knee. The IKDC Subjective Knee Form has been validated in Dutch and Italian as well as English.
Numeric Pain Rating Scale (NPRS) | 6 months
  The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme.
Goniometer: | 6 months
  The range of motion is the measurement of movement around a specific joint or body part. To measure the range of motion, doctors, osteopaths, physical therapists, or other health professionals most commonly use a goniometer, which is an instrument that measures angle motion at a joint.
Functional Strength Tests | 6 months
  Functionality testing following anterior cruciate ligament (ACL) reconstruction can benefit clinicians and patients in determining readiness for return to sport. The goals of testing following ACL reconstruction are to determine the strength of the muscles surrounding the knee, primarily the quadriceps and hamstrings, and evaluate knee stability and functionality through comparing the involved leg with the noninvolved leg.
  * Single Leg Hop
  * Test Single Leg Squat
  * Triple Hop Test
  * Treadmill
  * Cycling
  * Push up test (27)

CONTACTS AND LOCATIONS:
Overall Officials: Aamir Gul Memon, MS, Principal Investigator — Riphah International University
Locations (1):
- Bahawal Victoria Hospital, Bahawalpur, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Joreitz R, Lynch A, Rabuck S, Lynch B, Davin S, Irrgang J. PATIENT-SPECIFIC AND SURGERY-SPECIFIC FACTORS THAT AFFECT RETURN TO SPORT AFTER ACL RECONSTRUCTION. Int J Sports Phys Ther. 2016 Apr;11(2):264-78. PMID 27104060
- [Background] Cavanaugh JT, Saldivar A, Marx RG. Postoperative rehabilitation after posterior cruciate ligament reconstruction and combined posterior cruciate ligament reconstruction-posterior lateral corner surgery. Operative Techniques in Sports Medicine. 2015;23(4):372-84.
- [Background] Nelson C, Rajan L, Day J, Hinton R, Bodendorfer BM. Postoperative Rehabilitation of Anterior Cruciate Ligament Reconstruction: A Systematic Review. Sports Med Arthrosc Rev. 2021 Jun 1;29(2):63-80. doi: 10.1097/JSA.0000000000000314. PMID 33972483
- [Background] Perriman A, Leahy E, Semciw AI. The Effect of Open- Versus Closed-Kinetic-Chain Exercises on Anterior Tibial Laxity, Strength, and Function Following Anterior Cruciate Ligament Reconstruction: A Systematic Review and Meta-analysis. J Orthop Sports Phys Ther. 2018 Jul;48(7):552-566. doi: 10.2519/jospt.2018.7656. Epub 2018 Apr 23. PMID 29685058
- [Background] Kronenberger JN. What is the effectiveness of neuromuscular training versus traditional strength training on restoration of knee function in the rehabilitation of non-operative or post-operative anterior cruciate ligament patients? A Systematic Review: Walsh University; 2018.
- [Background] Huang DD, Chen LH, Yu Z, Chen QJ, Lai JN, Li HH, Liu G. Effect of suspension training on neuromuscular function, postural control, and knee kinematics in anterior cruciate ligament reconstruction patients. World J Clin Cases. 2021 Apr 6;9(10):2247-2258. doi: 10.12998/wjcc.v9.i10.2247. PMID 33869600
- [Background] Wang K, Cheng L, Wang B, He B. Effect of isokinetic muscle strength training on knee muscle strength, proprioception, and balance ability in athletes with anterior cruciate ligament reconstruction: a randomised control trial. Front Physiol. 2023 Sep 19;14:1237497. doi: 10.3389/fphys.2023.1237497. eCollection 2023. PMID 37795267
- [Background] Moubarak EES, Yousef EF, Dawood RS, El Shamy ASAH, Abdelrahem MEA. Effect of Adding Preoperative Exercise to Postoperative Rehabilitation Program of Progressive Exercises on Anterior Cruciate Ligament Reconstruction. Egyptian Journal of Physical Therapy. 2023;15(1):18-26.
- [Background] Walters SL. EFFECTS OF ACL RECONSTRUCTION ON MUSCULAR STRENGTH, ENDURANCE AND MITOCHONDRIAL CAPACITY: University of Georgia.
- [Background] Sigit M, Doewes M, Liskustyawati H. The effect of open kinetic chain exercise and close kinetic chain exercise on strength quadriceps femoris muscle post anterior cruciate ligament surgery in terms of age. Advances in Health and Exercise. 2024;4(1):10-6.
- [Background] Pamboris GM, Pavlou K, Paraskevopoulos E, Mohagheghi AA. Effect of open vs. closed kinetic chain exercises in ACL rehabilitation on knee joint pain, laxity, extensor muscles strength, and function: a systematic review with meta-analysis. Front Sports Act Living. 2024 Jun 3;6:1416690. doi: 10.3389/fspor.2024.1416690. eCollection 2024. PMID 38887689
- [Background] Qiu M. Comparison of Modalities and Strength and Motor Control Training Methods after Anterior Cruciate Ligament Reconstruction Surgery and Recommendations. MedScien. 2024;1(7).
- [Background] Gandhi KM, Ratnani G, Deodhe NP, Shende K. Enhancing Muscle Strength Post Anterior Cruciate Ligament Reconstruction: A Case Report Assessing the Effectiveness of Russian Current. Cureus. 2024 Feb 21;16(2):e54593. doi: 10.7759/cureus.54593. eCollection 2024 Feb. PMID 38524050
- [Background] Buckthorpe M. Optimising the Late-Stage Rehabilitation and Return-to-Sport Training and Testing Process After ACL Reconstruction. Sports Med. 2019 Jul;49(7):1043-1058. doi: 10.1007/s40279-019-01102-z. PMID 31004279
- [Background] Crank C, MOMT TMP. Rehabilitation Following Anterior Cruciate Ligament and Posterolateral Corner Reconstruction with Medial and Lateral Meniscus Repairs in A High School Athlete: A Retrospective Case Report. Orthopaedic Physical Therapy Practice. 2020;32(2):76-81.
- [Background] Welling W, Benjaminse A, Lemmink K, Dingenen B, Gokeler A. Progressive strength training restores quadriceps and hamstring muscle strength within 7 months after ACL reconstruction in amateur male soccer players. Phys Ther Sport. 2019 Nov;40:10-18. doi: 10.1016/j.ptsp.2019.08.004. Epub 2019 Aug 9. PMID 31425918
- [Background] Joreitz R, Lynch A, Popchak A, Irrgang J. CRITERION-BASED REHABILITATION PROGRAM WITH RETURN TO SPORT TESTING FOLLOWING ACL RECONSTRUCTION: A CASE SERIES. Int J Sports Phys Ther. 2020 Dec;15(6):1151-1173. doi: 10.26603/ijspt20201151. PMID 33344032
- [Background] Herman ZJ, Reddy RP, Fails A, Lin A, Popchak A. Rehabilitation and Return to Sport following Operative and Nonoperative Treatment of Anterior Shoulder Instability. Clin Sports Med. 2024 Oct;43(4):705-722. doi: 10.1016/j.csm.2024.03.025. Epub 2024 Apr 23. PMID 39232575
- [Background] Simonsson R, Piussi R, Hogberg J, Sundberg A, Hamrin Senorski E. Rehabilitation and Return to Sport After Anterior Cruciate Ligament Reconstruction. Clin Sports Med. 2024 Jul;43(3):513-533. doi: 10.1016/j.csm.2023.07.004. Epub 2023 Aug 23. PMID 38811125
- [Background] Ashoury H, Yalfani A, Arjipour M. The effects of open/closed kinetic chain exercises in water on the electrical activity of selected lumbar muscles, lumbopelvic control, ground reaction force and psychological factors in men with chronic non-specific low back pain: A study protocol for a randomized clinical trial. J Bodyw Mov Ther. 2024 Oct;40:2147-2154. doi: 10.1016/j.jbmt.2024.10.065. Epub 2024 Oct 25. PMID 39593577
- [Background] Forelli F, Mazeas J, Zeghoudi Y, Vandebrouck A, Duffiet P, Ratte L, Kakavas G, Hewett TE, Korakakis V, Rambaud AJM. Intrinsic graft laxity variation with open kinetic chain exercise after anterior cruciate ligament reconstruction: A non-randomized controlled study. Phys Ther Sport. 2024 Mar;66:61-66. doi: 10.1016/j.ptsp.2024.01.009. Epub 2024 Feb 6. PMID 38335650
- [Background] Girdwood M, Culvenor AG, Patterson B, Haberfield M, Rio EK, Hedger M, Crossley KM. No sign of weakness: a systematic review and meta-analysis of hip and calf muscle strength after anterior cruciate ligament injury. Br J Sports Med. 2024 Apr 25;58(9):500-510. doi: 10.1136/bjsports-2023-107536. PMID 38537939
- [Background] Trabka R, Maicki T, Kaminski P, Pawelczyk A, Zielinski P, Wilk-Franczuk M. Outcomes Following Arthroscopic Single and Double Bundle Anterior Cruciate Ligament (ACL) Reconstruction Supported by the Comprehensive Early Rehabilitation Program (CERP). Med Sci Monit. 2020 May 12;26:e921003. doi: 10.12659/MSM.921003. PMID 32396534
- [Background] Λιγνού Ε-Ά. Prevalence of central sensitizationsymptomsand psychosocial factors in athletes after ACL reconstruction and return to play 2020.
- [Background] HEDYA WM. Effect of different exercise rehabilitation programs with body weight reduction on reducing the time of injured limb efficient restoration before and after low knee osteotomy surgery. International Journal of Sports Science and Arts. 2019;4(04):59-78.
- [Background] Lopez-Valenciano A, Ayala F, De Ste Croix M, Barbado D, Vera-Garcia FJ. Different neuromuscular parameters influence dynamic balance in male and female football players. Knee Surg Sports Traumatol Arthrosc. 2019 Mar;27(3):962-970. doi: 10.1007/s00167-018-5088-y. Epub 2018 Aug 7. PMID 30088029
- [Background] Buckthorpe M, La Rosa G, Villa FD. RESTORING KNEE EXTENSOR STRENGTH AFTER ANTERIOR CRUCIATE LIGAMENT RECONSTRUCTION: A CLINICAL COMMENTARY. Int J Sports Phys Ther. 2019 Feb;14(1):159-172. PMID 30746302
- [Background] Mayer MA, Deliso M, Hong IS, Saltzman BM, Longobardi RS, DeLuca PF, Rizio L. Rehabilitation and Return to Play Protocols After Anterior Cruciate Ligament Reconstruction in Soccer Players: A Systematic Review. Am J Sports Med. 2025 Jan;53(1):217-227. doi: 10.1177/03635465241233161. Epub 2024 Apr 15. PMID 38622858
- [Background] Taş B, Ok E, Akalp U, Bingül BM, Gelen E. Effect of lower extremity joint distraction exercises during warm-up on range of motion, flexibility, and jump performance in female volleyball players. Pedagogy of Physical Culture and Sports. 2024;28(4):283-91.
- [Background] Sievert ZA. The Effects of Anterior Cruciate Ligament Thickness, Knee Joint Laxity, Activity Level, Neuromuscular Imbalances and Lower Extremity Muscular Activation Patterns on Anterior Cruciate Ligament Loading: Old Dominion University; 2019.
- [Background] Peel SA, Schroeder LE, Weinhandl JT. Lower extremity muscle contributions to ACL loading during a stop-jump task. J Biomech. 2021 May 24;121:110426. doi: 10.1016/j.jbiomech.2021.110426. Epub 2021 Apr 9. PMID 33873112
- [Background] Piskin D, Benjaminse A, Dimitrakis P, Gokeler A. Neurocognitive and Neurophysiological Functions Related to ACL Injury: A Framework for Neurocognitive Approaches in Rehabilitation and Return-to-Sports Tests. Sports Health. 2022 Jul-Aug;14(4):549-555. doi: 10.1177/19417381211029265. Epub 2021 Jul 8. PMID 34236003
- [Background] Bram JT, Magee LC, Mehta NN, Patel NM, Ganley TJ. Anterior Cruciate Ligament Injury Incidence in Adolescent Athletes: A Systematic Review and Meta-analysis. Am J Sports Med. 2021 Jun;49(7):1962-1972. doi: 10.1177/0363546520959619. Epub 2020 Oct 22. PMID 33090889
- [Background] Bloom DA, Wolfert AJ, Michalowitz A, Jazrawi LM, Carter CW. ACL Injuries Aren't Just for Girls: The Role of Age in Predicting Pediatric ACL Injury. Sports Health. 2020 Nov/Dec;12(6):559-563. doi: 10.1177/1941738120935429. Epub 2020 Aug 11. PMID 32780637
- [Background] Colombo V, Valencic T, Steiner K, Skarabot J, Folland J, O'Sullivan O, Kluzek S. Comparison of Blood Flow Restriction Interventions to Standard Rehabilitation After an Anterior Cruciate Ligament Injury: A Systematic Review. Am J Sports Med. 2024 Dec;52(14):3641-3650. doi: 10.1177/03635465241232002. Epub 2024 Apr 9. PMID 38591459
- [Background] Ong MT, Chan JS, Man GC, Qiu J, He X, Wang Q, Yung PS. Effect of eccentric isokinetic exercise on muscle strength and functional recovery after anterior cruciate ligament reconstruction. Asia Pac J Sports Med Arthrosc Rehabil Technol. 2023 Nov 24;35:20-26. doi: 10.1016/j.asmart.2023.11.002. eCollection 2024 Jan. PMID 38075532
- [Background] Wong CT, Mok KM, Yung SP. Secondary Anterior Cruciate Ligament Injury Prevention Training in Athletes: What Is the Missing Link? Int J Environ Res Public Health. 2023 Mar 9;20(6):4821. doi: 10.3390/ijerph20064821. PMID 36981735
- [Background] Piussi R, Krupic F, Senorski C, Svantesson E, Sundemo D, Johnson U, Hamrin Senorski E. Psychological impairments after ACL injury - Do we know what we are addressing? Experiences from sports physical therapists. Scand J Med Sci Sports. 2021 Jul;31(7):1508-1517. doi: 10.1111/sms.13959. Epub 2021 Apr 6. PMID 33772890